CLINICAL TRIAL: NCT03975062
Title: "Prospective Open Label Randomized Evaluation of Abbreviated Course of Dabigatran Etexilate With tranSesophageal echOcardiography (TEE) Control vs Conventional 3-week coUrse With dabigatraN Etexilate Before Cardioversion: Analysis of MRI-detecteD Cerebral Embolism" (RE-SOUND Study), № 1160.242
Brief Title: Evaluation of Abbreviated Versus Conventional Course of Dabigatran Etexilate Before Electric Cardioversion in Patients With Atrial Fibrillation (RE-SOUND Study)
Acronym: RE-SOUND
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ural State Medical University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Vadim Grachev, Principal Investigator, Ural State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1160.242
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cardioversion; anticoagulation; dabigatran; magnetic resonance imaging
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Intervention Model Description: PROBE design, multicenter, active control trial
Who Masked: Outcomes Assessor
Masking Description: Blinded evaluation of primary outcome by Imaging expert, who will made decision regarding achievement of primary outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abbreviated course group (ACG) (Experimental): The patients receiving 3-days course of dabigatran etexilate during pre-cardioversion period. After cardioversion has been performed the patients continue with dabigatran etexilate until 30 days after cardioversion
  Interventions: Drug: dabigatran etexilate
- Conventional course group (CCG) (Active Comparator): The patients receiving 3-weeks course of dabigatran etexilate before cardioversion of AF. After cardioversion has been performed the patients will continue with dabigatran etexilate until 30 days after cardioversion
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — 150 mg twice daily (BID)

SUMMARY:
The purpose of the study is to evaluate the efficacy of abbreviated 3-day anticoagulation with dabigatran etexilate before cardioversion guided by trans-oesophageal echocardiography in comparison with conventional 3- week course of dabigatran etexilate before cardioversion

DETAILED DESCRIPTION:
Current guidelines recommend for stroke prevention in patients with atrial fibrillation (AF) lasting more than 48 h designated for cardioversion standard approach with anticoagulation for a minimum 3 weeks before anticoagulation. The alternative is abbreviated anticoagulation in case of using trans-oesophageal echocardiography (TEE)-guided approach with quick cardioversion if no thrombus or high-grade spontaneous echo contrast is seen. There is currently no data on the direct comparison of efficacy and safety of conventional and abbreviated courses of non-vitamin K antagonist oral anticoagulants (NOAC) before cardioversion in AF.

The RE-SOUND study is prospective open label study with blinded outcome evaluation (PROBE design) multicenter active control trial comparing efficacy of 3-day abbreviated TEE-guided and conventional 3-week courses of NOAC dabigatran etexilate before cardioversion in adult patients with AF lasting more than 48 h

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged >18 years old and <75 years old
* the diagnosis of non-valvular atrial fibrillation/atrial flutter duration of 48 hours or more (or unknown) documented by ECG. Duration of AF will be defined on the base of patient source documents
* documented physician's decision to conduct electrical cardioversion
* written informed consent form (ICF) signed by patient

Exclusion Criteria:

* effective treatment with oral anticoagulants within the last 30 days
* need in anticoagulant treatment for disorder other than AF
* rheumatic heart disease
* mitral stenosis of unknown origin
* mechanic heart valve
* acute coronary syndrome within 12 months
* percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery within the last 12 month or planned for the next 8 weeks
* known hypersensitivity for dabigatran, dabigatran etexilate or to any of capsul's components
* creatinine clearance <30 ml/min
* active bleeding, haemorrhagic diathesis, coagulopathy
* major surgery within the previous month, surgery planned for the next 8 weeks,
* clinically relevant bleeding within the last 30 days
* symptomatic or endoscopically documented gastroduodenal ulcers within the last 30 days
* intracranial haemorrhages in medical history
* organ damages resulted from clinically relevant bleeding within 6 months before randomization.
* major trauma or any craniocerebral trauma within 30 days before randomization.
* any cancer within last 5 years
* uncontrolled hypertension (systolic blood pressure >180mm Hg and/or diastolic blood pressure >100 mmHg).
* chronic heart failure (CHF) III-IV functional classes (by NYHA)
* severe ischemic stroke within the last 12 month before randomization
* changes of liver functions with alanine aminotransferase (ALT)/aspartate aminotransferase (AST) >3 upper limit of normal (ULN)
* liver disease having impact on survival
* pregnancy and breast feeding. Women of child bearing potential must agree to the requirements for pregnancy testing and contraceptive methods
* any contraindications for electric cardioversion (see attachment # 1 for details).
* any contraindications to cerebral MRI
* any contraindications to TEE ( perforated viscus; esophageal pathology (stricture, trauma, tumor, scleroderma, Mallory-Weiss tear, diverticulum); tracheoesophageal fistula; active upper GI bleeding; recent upper GI surgery; esophagectomy, esophagogastrectomy.)
* patients who on the discretion of physician will not benefit from 150 BID dose of dabigatran during study course
* active hepatitis
* anemia (hemoglobin level <100g/L) or thrombocytopenia (platelet count <100 × 109/L)
* alcohol abuse
* hyperthyroidism

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with new magnetic resonance imaging (MRI) detected cerebral embolic events | 30 days after cardioversion
  patients with new (not visible at pre-cardioversion MRI) cerebral ischemic lesions revealed at MRI after cardioversion and without a history of acute neurological dysfunction attributable to the lesion or with symptomatic cerebral ischemic stroke after cardioversion confirmed by MRI examination

SECONDARY OUTCOMES:
the incidence of symptomatic cerebral thromboembolic events (stroke or TIA) | within 30 days after cardioversion
  An acute episode of focal or global neurological dysfunction caused by brain, spinal cord or retinal vascular injury as a result of hemorrhage or infarction (with imaging, pathological or other objective evidence of cerebral, spinal cord or retinal injury or clinical evidence with symptoms persisting ≥24 hours or until death and other etiology excluded) or transient (<24 hours) episode of focal neurological dysfunction caused by brain, spinal cord or retinal ischemia without acute infarction
the proportion of patients with major bleeding events after cardioversion | within 30 days after cardioversion
  major bleeding as defined by the International Society of Thrombosis and Hemostasis (ISTH) criteria
the proportion of patients with any bleeding events after cardioversion | within 30 days after cardioversion
  any clinical obvious bleeding
the proportion of patients with intracranial bleeding events after cardioversion | within 30 days after cardioversion
  symptomatic intraparenchymal, intraventricular, subarachnoid, subdural, epidural hemorrhage with imaging or pathological evidence
the proportion of patients with at least one bleeding event since the first dose of dabigatran | from the first dose of dabigatran etexilate till 30th day after cardioversion
  any clinical obvious bleeding
the proportion of patients with at least one major bleeding event since the first dose of dabigatran | from the first dose of dabigatran etexilate till 30th day after cardioversion
  major bleeding as defined by the ISTH criteria
the proportion of patients with intracranial bleeding events since the first dose of dabigatran | from the first dose of dabigatran etexilate till 30th day after cardioversion
  symptomatic intraparenchymal, intraventricular, subarachnoid, subdural, epidural hemorrhage with imaging or pathological evidence

OTHER OUTCOMES:
rate of sinus rhythm restoration after cardioversion | within 30 days after cardioversion
  achieving and maintaining of sinus rhythm for at least 10 min after shock
rate of AF recurrence | from 10 minutes till 30th day after cardioversion
  recurrent episodes of AF or atrial flutter
the time until restoration of left atrial (LA) mechanic function | during 5 days from cardioversion until peak A revealed or until atrial fibrillation recurrence (if this happens before)
  transmitral flow peak A restoration on results of echocardiography
D-dimer concentration | at the time of cardioversion, 1 day after cardioversion and 10 days after cardioversion
  D-dimer concentration in laboratory evaluation in sub-set of 100 patients only at one pre-selected investigational site
brain natriuretic peptide (BNP) level | right before cardioversion
  BNP level in laboratory evaluation in sub-set of 100 patients only at one pre-selected investigational site
E/E' ratio | before cardioversion
  the ratio of transmitral Doppler early filling velocity to tissue Doppler early diastolic mitral annular velocity on results of echocardiography
flow velocity in the left atrial appendage (LAA) | precardioversion day
  flow velocity in the LAA TEE evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Olga G Smolenskaya, MD, Study Chair — Ural State Medical University; Vadim G Grachev, PhD, Principal Investigator — Ural State Medical University
Locations (1):
- Limited Liability Company Medical Association "Novaya Bolnitsa", Yekaterinburg, Russia

IPD SHARING:
Plan to Share IPD: No